CLINICAL TRIAL: NCT05001893
Title: Clinical Safety and Efficacy of S53P4 Bioactive Glass Putty in Spinal Fusion Surgery: Post Market Clinical Follow-up Study
Brief Title: Clinical Safety and Efficacy of S53P4 Bioactive Glass Putty in Spinal Fusion Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Bonalive Biomaterials Ltd (Industry)
Collaborators: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 103-CL01
Record Dates: First submitted 2021-05-04; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-07

CONDITIONS: Spine Fusion; Spinal Deformity
Keywords: S53P4; Bonalive; Bioactive glass putty; Spine fusion; Lumbar spine fusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The use of a mixture of BonAlive® putty and autologous bone: A retrospective case-controlled study will be created to compare the use of a mixture of BonAlive® putty and autologous bone to autologous bone alone for clinical safety and efficacy.
  Interventions: Device: S53P4 bioactive glass putty

INTERVENTIONS:
Device: S53P4 bioactive glass putty — Bonalive putty/putty MIS paste is a synthetic, bioactive, osteoconductive, osteostimulative bone void filler for filling, reconstruction, and regeneration of bone defects.
  Other Names: Bonalive® putty, Bonalive® putty MIS

SUMMARY:
A retrospective, single-tertiary centre observational study.

The study population consists mainly of patients with instrumented posterolateral spine fusion operated at the Department of Neurosurgery or at the Department of Orthopaedics and Traumatology in the Turku University Hospital. Also, patients with non-instrumented posterolateral spine fusion, interbody spine fusion, and a combination of posterolateral and interbody spine fusion are included.

The approximate number of the above-mentioned operations with BonAlive® putty is 400 - 500 between September 2013 and April 2021. In the operations, the BonAlive® putty was used either alone, together with autologous bone (AB) chips, with milled allogenous bone chips, with demineralized bone matrix (DBM), with other synthetic bone grafts, or with a combination of the above-mentioned.

DETAILED DESCRIPTION:
In the first stage of the investigation, the clinical safety and efficacy of BonAlive® putty are assessed in a retrospective case-series, and the observations are compared to the existing literature. Thereafter, a retrospective case-controlled study will be created to compare the use of a mixture of BonAlive® putty and AB to AB alone for clinical safety and efficacy. The cases will be matched up with the controls by gender, age, smoking behavior, the number of operated levels and the site of operated levels as far as possible. The chosen surgical technique will be the most commonly used.

ELIGIBILITY:
Inclusion Criteria:

1. Performed spine fusion operation
2. BonAlive® putty used in the operation

Exclusion Criteria:

1. Age under 18
2. Use of other synthetic bone graft substitute or expander materials than BonAlive® putty in the operation
3. Less time than two years since the index operation and no CT-proof of intended bony fusion

Age Groups: Child, Adult, Older Adult
Study Population: The study population consists mainly of patients with instrumented posterolateral spine fusion operated at the Department of Neurosurgery or at the Department of Orthopaedics and Traumatology in the Turku University Hospital. Also, patients with non-instrumented posterolateral spine fusion, interbody spine fusion, and a combination of posterolateral and interbody spine fusion are included.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the clinical efficacy of BonAlive® (S53P4 bioactive glass) putty in spine fusion operations when used alone and together with autologous bone. | 24 months
  Radiologic endpoints are based on a neuroradiologist evaluatyion possible complications (breakage and/or loosening of the instrumentation) and bony fusion on a modified Bridwell grading criteria I-IV for PLF.
Clinical outcomes are for pain VAS: | 24 months
  Visual analogue scale 1-10.
EQ-5D cost effectiviness questionnaires. | 24 months
  Values are anchored at 1 (full health) and 0 (a state as bad as being dead) as required by their use in economic evaluation.
ODI: (Oswestry Low Back Pain Disability Questionnaire). | 24 months
  ODI is validated to use in patients with low back pain.The final score/index ranges from 0-100. A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound.
15 D questionnaire The 15D is a generic, comprehensive (15-dimensional), self-administered instrument for measuring HRQoL among adults. | 24 months
  Health index on a 0-1 scale has been used successfully in several pharmacoeconomic evaluations. The maximum score is 1 (no problems on any dimension) and the minimum score is 0 (being dead).

SECONDARY OUTCOMES:
To demonstrate that the clinical efficacy of BonAlive® putty used together with autologous bone in spine fusion operations is not inferior to the clinical efficacy of autologous bone used alone. | 24 months
  Radiologic endpoints are based on a neuroradiologist evaluation possible complications; 1. breakage and/or loosening of the instrumentation 2. bony fusion on a modified Bridwell grading criteria for PLF.
To demonstrate that the clinical use of BonAlive® putty does not cause excess infections or other complications subsequent to spine fusion operations compared to the reported amounts in the literature without the use of BonAlive® putty. | 24 months
  Odom´s scale
  1 Excellent: No symptoms related to cervicaldisease.Able to perform daily activities without limitations. 2 Good: Moderate symptoms related tocervical disease.Able to perform daily activities without significant limitations. 3 Satisfactory: Slight improvement in symptomsrelated to cervical disease.Significant limitations in daily activities. 4 Poor: No improvement in, or aggravation of,symptoms related to cervical disease.Not able to perform daily activities.

OTHER OUTCOMES:
• To demonstrate that the clinical use of BonAlive® putty does not cause excess infections or other complications subsequent to spine fusion operations compared to the reported amounts in the literature without the use of BonAlive® putty. | 24 months
  Re-operations and infections in the area of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ilkka Saarenpää, MD, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital Department of Neurosurgery, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided